CLINICAL TRIAL: NCT05357495
Title: Characterization and Pathophysiology of Frustration in Pediatric Irritability
Brief Title: Characterization and Brain Mechanisms of Frustration in Youth With Severe Irritability or Attention Deficit Hyperactivity Disorder (ADHD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is retiring
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10000774; 000774-M
Record Dates: First submitted 2022-04-29; First posted 2022-05-03 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Disruptive Mood Dysregulation Disorder; Attention Deficit Hyperactivity Disorder; Normal Physiology
Keywords: Magnetic Resonance Imaging; Resting State; Task Based
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- frustration and control fMRI tasks (Experimental): all subjects complete one scanning session with frustration induction and one scanning session with the control task.
  Interventions: Behavioral: Affective Posner fMRI frustration induction task

INTERVENTIONS:
Behavioral: Affective Posner fMRI frustration induction task — During the frustration induction paradigm, children play a game with monetary reward. The game is rigged, thus inducing frustration. The control task does not have any reward component. All participants complete both the control task scanning session and the frustration induction scanning session.

SUMMARY:
Background:

Irritability is an elevated proneness to anger. Children with irritability have difficulty tolerating frustration. They get angry and have temper outbursts more easily than their others their age. Irritability is a symptom of DMDD and ADHD. (DMDD is disruptive mood dysregulation disorder. ADHD is attention deficit/hyperactivity disorder.) Yet the reasons why some children get irritated easily are not well understood.

Objective:

To use brain imaging methods to study responses to frustration in youth.

Eligibility:

Youth aged 8 to 17 years with severe irritability (including those diagnosed with DMDD) and/or ADHD. Healthy volunteers are also needed. All participants are already enrolled in studies 02-M-0021 or 01-M-0192.

Design:

Participants will visit the clinic 3 times. The second and third visits will be 3 to 4 weeks apart.

The first visit will be an enrollment visit. They will receive training on the tasks they will do during the study. Participants and their parents will take surveys. They will answer questions about their moods and feelings.

Participants will train for an MRI scan. They will lie in a mock scanner tube and hear the noises an MRI makes.

On the second and third visits, participants will have real MRI scans. They will play a computer game or watch a movie during each scan. The scans will last about 1 hour.

The week after each scan, participants will wear a device on their wrist to measure their heart rate and activity level. Participants and their parent will use a smartphone to answer questions about how they are feeling and acting. Participants who do not have smartphones will be given one to use during the study.

DETAILED DESCRIPTION:
Study Description:

Participants in this study will be drawn from those enrolled in Protocol 02-M-0021 or 01-M-0192. This protocol uses detailed clinical phenotyping and a frustration induction task, coupled with pre- and post-frustration resting state scans, to study brain mechanisms mediating severe irritability in youth. The primary objective is to identify brain networks contributing to reconfiguration during and after frustration, and to test the ability of brain network metrics obtained using a frustration induction task to predict irritability. The secondary objective is to test whether these predictions are strengthened by the addition of structural connectivity measures and deeper clinical phenotyping.

Objectives:

Primary Objective:

To use multi-modal functional magnetic resonance imaging (fMRI), including a frustration induction task, coupled with resting state functional connectivity (rsFC) pre- and post-frustration, to elucidate neural mechanisms mediating frustration and how aberrant responses to frustration contribute to severe irritability in youth. Specifically, we will identify brain networks contributing to reconfiguration during and after frustration and test the ability of brain network metrics to predict irritability.

Secondary Objectives:

To test whether the prediction of irritability can be improved by the addition of structural brain connectivity measures obtained using diffusion tensor imaging (DTI), and clinical measures i.e., real-time, ecologically valid measures of mood and behavior obtained using ecological momentary assessment (EMA).

Endpoints:

Primary Endpoints:

Global efficiency (Eglob) of brain modules during resting state after frustration, which we hypothesize will predict irritability. Variance of information (VIn) measures, which we hypothesize will demonstrate that anterior DMN-temporal-limbic (aDMN-TL) and fronto-parietal (FP) modules make the largest contributions to network reconfiguration throughout frustration.

Secondary Endpoints:

Measures of structural connectivity obtained using DTI, and EMA measures of mood and behavior, which we hypothesize will improve the prediction of irritability.

ELIGIBILITY:
* INCLUSION CRITERIA:

This study will include patients (i.e., youth with DMDD subthreshold DMDD, and/or ADHD) and healthy volunteers. All subjects will have already been enrolled in 02-M-0021 or 01-M-0192.

Inclusion criteria for patients:

* Enrolled in 02-M-0021.
* Aged 8-17 at the time of recruitment.

Healthy Volunteer Children

* Enrolled in 02-M-0021 or 01-M-0192 as a healthy volunteer.
* Aged 8-17 at the time of recruitment.

EXCLUSION CRITERIA:

-An individual who has contraindications for scanning will be excluded.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
prediction of irritability ratings by global efficiency | one week after each of two scanning sessions, when ecological momentary assessment ratings are completed. The two scanning sessions will be 2-5 weeks apart.
  global efficiency of brain modules in resting state after frustration will be used to predict irritability ratings obtained throughout the one week after each of two scanning sessions
Variance of information (VIn) measures | data are obtained throughout each of the two scanning sessions. The two scanning sessions will be 2-5 weeks apart.
  VIn metric will be used to identify the brain modules making the largest contribution to network reconfiguration throughout frustration

SECONDARY OUTCOMES:
ecological momentary assessment (EMA) measures | for one week after each of the two scanning sessions
  Remote digital phenotyping will be used to assess mood and behavior throughout the week following each of the two scanning sessions. These EMA measures will be included in a machine learning model to test whether their inclusion can improve the prediction of irritability ratings.
Diffusion tensor imaging (DTI) metrics | during first scanning session
  Standard DTI metrics will be included in a machine learning model to test whether their inclusion can improve the prediction of irritability ratings.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Leibenluft, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Starting six months after publication and ending five years later
Access Criteria: All data will be available that are allowable based on IRB-approved procedures.(SqrRoot)

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000774-M.html